CLINICAL TRIAL: NCT01469858
Title: Perception and Multisensory Integration in Neurological Patients Using fMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 044811HMO
Record Dates: First submitted 2011-11-01; First posted 2011-11-10 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-09

CONDITIONS: Acute Inflammatory Demyelinating Polyradiculoneuropathy; Myasthenia Gravis; Stroke; Anosognosia; Asomatognosia
MeSH Terms: conditions — Guillain-Barre Syndrome; Myasthenia Gravis; Stroke; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study group (Experimental): fMRI
  Interventions: Device: Siemens magnetom avanto1.5 Tesla, Siemens magnetom trio A Tim system 3 Tesla

INTERVENTIONS:
Device: Siemens magnetom avanto1.5 Tesla, Siemens magnetom trio A Tim system 3 Tesla — functional magnetic resonance imaging

SUMMARY:
The main objective of the study is to explore and map brain areas involved in sensory perception and multisensory integration in patients with central or peripheral neurological damage. The investigators hypothesize for example, that a change (compare to healthy subjects) in the perceptual maps and body representation could be detected and characterize in patients suffering from impairments of peripheral nerve conduction.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of the investigated neuronal disease

Exclusion Criteria:

* contraindication for MRI scan
* pregnancy
* refusal to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
assessing hemodynamic responses by measurement of the Blood-oxygen-level dependence(BOLD)signal | 1 year
  Distinct maps of sensory and multisensory representations related to certain disorders will be assed by measurement of the Blood-oxygen-level dependence(BOLD)signal.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Arzy S, Overney LS, Landis T, Blanke O. Neural mechanisms of embodiment: asomatognosia due to premotor cortex damage. Arch Neurol. 2006 Jul;63(7):1022-5. doi: 10.1001/archneur.63.7.1022. PMID 16831974